CLINICAL TRIAL: NCT02233140
Title: Do Physical Manipulation Exercises With EPAT Improve Ankle Dorsiflexion and Reduce Dynamic Plantar Forefoot Pressure in Diabetic Subjects With Equinus?: A Pilot RCT
Brief Title: Effectiveness of Manual Manipulation With EPAT on Ankle Dorsiflexion and Dynamic Plantar Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21660
Record Dates: First submitted 2014-08-28; First posted 2014-09-08 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes; Equinus Contracture of the Ankle
Keywords: Diabetes; Ankle equinus; ankle dorsiflexion; dynamic plantar pressure; shockwave therapy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shockwave with manual manipulation (Experimental): A shockwave (EPAT) therapy with two supervised manual manipulation per week
  Interventions: Device: Extra-corporeal pulsed-activated therapy or shockwave therapy
- Manual manipulation (Active Comparator): A Placebo (no) shockwave with two supervised manual manipulations per week
  Interventions: Device: Extra-corporeal pulsed-activated therapy or shockwave therapy

INTERVENTIONS:
Device: Extra-corporeal pulsed-activated therapy or shockwave therapy
  Other Names: D-Actor® 200

SUMMARY:
Diabetic foot complications are a common and costly problem. Excessive plantar pressures due to foot deformities and/or limited ankle dorsiflexion, especially in the presence of peripheral neuropathy, can predispose subjects with diabetes for diabetic foot ulcers. Achilles tendon lengthening surgery has shown to delay or prevent recurrence of diabetic foot ulcers.

Studies have shown that Shockwave Therapy (EPAT - Extracorporeal Pulse Activation Technology) was effective in treating subjects with chronic heel pain and Achilles tendonitis with no serious side effects. EPAT, therefore, may allow diabetic patients with ankle equinus to perform more effective stretching exercises and may prevent recurrence of diabetic foot ulcers.

The purposed of this RCT is to compare effectiveness of manual manipulation with EPAT versus manual manipulation alone on ankle dorsiflexion and dynamic plantar pressure in at-risk subjects with a history of diabetic foot ulcer.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 21 to 65, inclusive
* Diabetes, either type 1 or 2
* Ankle equinus (< 0º passive ankle dorsiflexion with knee extended)
* Forefoot plantar hyperkeratosis (callus)
* Able to walk independently without the use of walking aids (cane, crutches, or walker)
* Able to understand the information in the informed consent form and willing and able to comply with study-related procedures

Exclusion Criteria:

* Previous history of ankle-foot surgery or amputation
* no active lower extremity skin ulcers
* Peripheral vascular disease (non-palpable pedal pulses or ankle brachial index <0.8)
* Not willing or able to make required visits
* Nursing or pregnant
* Not willing or able to follow procedures specified by protocol and/or instructions of the study personnel, including discontinuation of icing, NSAIDs and natural anti-inflammatory agents (such as Arnica)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Change in maximum ankle dorsiflexion (lunge test) from baseline to 4 weeks | at baseline visit and at 4 weeks
Change in dynamic peak plantar pressure (sub-metatarsal 2) in barefoot walking from baseline to 4 weeks. | at baseline visit and 4 weeks

SECONDARY OUTCOMES:
Change in maximum ankle dorsiflexion (lunge test) from 1 month to 3 months. | at 1 month and at 3 months
Change in dynamic peak plantar pressure (sub-metatarsal 2) in barefoot walking from 1 month to 3 months. | at 1 month and at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jinsup Song, DPM, PhD, Principal Investigator — Temple University
Locations (1):
- Gait Study Center at the Temple University School of Podiatric Medicine, Philadelphia, Pennsylvania, United States